CLINICAL TRIAL: NCT06847958
Title: HepC Micro-elimination on MSM Comunity
Brief Title: HepC Micro-elimination on MSM and TGW Population.
Status: Completed | Type: Observational
Sponsor: Projecte dels NOMS Hispanosida (Other)
Collaborators: Fundació Lluita contra les Infeccions (Unknown); Germans Trias i Pujol Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MSM-HCV-MicroElimination; IN-ES-987-5997 (Other Grant/Funding Number: Gilead Sciences, S.L.U); PI-21-206 (Registry Identifier: IEC Germans Trias i Pujol)
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Hepatitis C; PrEP; Drugs of Abuse
Keywords: MSM; TGW; PrEP; Hepatitis C Transmision; micro-elimination
MeSH Terms: conditions — Hepatitis C; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MSM and TGW HIV negative PrEP User.
- MSM and TGW HIV negative non PrEP User.

SUMMARY:
This is an observational study, in which a single visit will be carried out, which includes a questionnaire on sexual habits and in which the possibility of carrying out a screening for Hepatitis C will be offered. Depending on the score obtained in the questionnaire, the screening will be carried out using a rapid serology test or viral load. During the first year, a SCORE will be developed to classify the risk of positive results. This SCORE will be used during phase 2 to offer users of the centres a targeted screening based on the Pre-test score.

ELIGIBILITY:
Inclusion Criteria:

1. All BCN Checkpoint and BCN PreP·Point clients.
2. 18 years and older.
3. HIV uninfected or diagnosticated in the center in the last 7 days prior to the study inclusion.
4. Men that have sex with men or transgender women.
5. Signature of written consent form.
6. Ability to comply with the requirements of the study protocol.

Exclusion Criteria:

1. Knowledge of HIV infection from more than 7 days
2. Knowledge of active HCV infection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male and TGW
Study Population: Men who have sex with other men or transgender women, that are HIV negative and comes to get tested in our center or are under controls in our center. Estimated enrollment first Phase 6000-7000 participants. Second phase 2000-3000 participants.
Sampling Method: Non-Probability Sample
Enrollment: 13161 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Hepatitis C active infection | August 2021 o September 2023
  Confirmed Hepatitis C active infection

CONTACTS AND LOCATIONS:
Locations (1):
- BCN checkpoint, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data requisition will be individually evaluated. After that IEC will be required to evaluate data sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be availeble up to 5 years after Data publication
Access Criteria: Data acces under private requisition and after individual evaluation.

REFERENCES:
- [Derived] Rivero A, Dalmau-Bueno A, Perez F, Coll P, Cabrera JM, Lucejko M, Fernandez J, Reguant J, Calderon J, Romero J, Caballero F, Marazzi G, Oro C, Michael Jacobs D, Vicioso H, Moises L, Taboada H, Saz J, Pujol F, Meulbroek M, Paredes R. HCV infection, risk factors and PrEP use among HIV-negative MSM and TW at a community health centre. J Infect Public Health. 2026 Feb;19(2):103086. doi: 10.1016/j.jiph.2025.103086. Epub 2025 Dec 4. PMID 41380408

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/58/NCT06847958/Prot_SAP_ICF_000.pdf